CLINICAL TRIAL: NCT00255554
Title: Effects of Dialectical Behavioral Therapy and Escitalopram on Impulsive Aggression, Affective Instability and Cognitive Processing in Borderline Personality Disorder
Brief Title: DBT and Escitalopram in Borderline Personality Disorder
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Bronx VA Medical Center (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 3277-03-0027
Record Dates: First submitted 2005-11-17; First posted 2005-11-21 (Estimated); Last update posted 2005-11-21 (Estimated); Status verified 2005-11

CONDITIONS: Borderline Personality Disorder
Keywords: Borderline Personality Disorder; BPD; Dialectical Behavior Therapy; DBT; Escitalopram; Lexapro
MeSH Terms: conditions — Borderline Personality Disorder | interventions — Escitalopram

INTERVENTIONS:
Behavioral: Dialectical Behavioral Therapy
Drug: Escitalopram

SUMMARY:
Subjects will receive six months of DBT, consisting of one 90-minute group and one 60-minute individual session per week as well as telephone availability of the individual therapist. Half the subjects will concurrently receive escitalopram while half will receive placebo, in a randomized double-blind design.

ELIGIBILITY:
Inclusion Criteria: Is a male or female between 18 and 60 who meets criteria for Borderline Personality Disorder and has been off psychotropic medications for at least 2 weeks (6 weeks for fluoxetine).

-

Exclusion Criteria: Meets criteria for Schizophrenia, Bipolar Disorder, Mental Retardation, current or recent Substance Dependence or a current Major Depressive Episode. Subjects also should not currently be in individual psychotherapy. (Case management and work therapy programs are allowed.)

-

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult

PRIMARY OUTCOMES:
Measures of impulsivity, aggression, affective impulsivity, immediate and delayed memory, and cognitive processing at baseline, 6 months and 9 months

CONTACTS AND LOCATIONS:
Overall Officials: Marianne Goodman, MD, Principal Investigator — Bronx VA Medical Center/Mount Sinai School of Medicine
Locations (1):
- Bronx VA Medical Center, The Bronx, New York, United States

REFERENCES:
- [Derived] Stoffers-Winterling JM, Storebo OJ, Pereira Ribeiro J, Kongerslev MT, Vollm BA, Mattivi JT, Faltinsen E, Todorovac A, Jorgensen MS, Callesen HE, Sales CP, Schaug JP, Simonsen E, Lieb K. Pharmacological interventions for people with borderline personality disorder. Cochrane Database Syst Rev. 2022 Nov 14;11(11):CD012956. doi: 10.1002/14651858.CD012956.pub2. PMID 36375174